CLINICAL TRIAL: NCT00211497
Title: A Phase II, Randomized, Vehicle-Controlled, Double-Blind, Multi-Center Study to Evaluate Safety and Efficacy of MBI 226 1.25% and 2.5% Acne Solutions Applied Topically for 12 Weeks to Subjects With Acne Vulgaris
Brief Title: Safety and Efficacy of MBI 226 1.25% and 2.5% Topical Acne Solutions in the Treatment of Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioWest Therapeutics Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A99005
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Acne Vulgaris; Acne; Propionibacterium Acnes
Keywords: acne vulgaris; acne; Propionibacterium acnes; topical; inflammatory; non-inflammatory; lesion counts; lesions
MeSH Terms: conditions — Acne Vulgaris

INTERVENTIONS:
Drug: MBI 226 Acne Solutions

SUMMARY:
This is a Phase II, randomized, vehicle-controlled, double-blind, multi center study to evaluate the efficacy and safety of topically applied MBI 226 1.25% and 2.5% Acne Solutions as anti-acne preparations in human subjects with facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 12 years and older
* Presence of inflammatory and non-inflammatory lesions

Exclusion Criteria:

* Acne conglobata, acne fulminans, or secondary acne (chloracne, drug-induced acne, etc.)
* Active facial cysts or any nodulocystic lesions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255
Dates: Start 2003-01; Study Completion 2003-09

PRIMARY OUTCOMES:
- percent change from Baseline to Week 12 in inflammatory acne lesion counts

SECONDARY OUTCOMES:
Single continuous endpoints:
• Percent change from Baseline to Week 6 and Week 12 in non inflammatory acne lesion counts
• The percent change from Baseline to Week 6 and Week 12 in total acne lesion counts
Multiple continuous endpoints:
• Percent change from Baseline to Weeks 3, 6, 9 and 12 in inflammatory acne lesion counts
• Percent change from Baseline to Weeks 3, 6, 9 and 12 in non-inflammatory acne lesion counts
• Percent change from Baseline to Weeks 3, 6, 9 and 12 in total acne lesion counts
Categorical endpoints:
• Dichotomized Physicians Global Severity Assessment scores at Week 6 and Week 12
• PGSA absolute scores at Week 6 and Week 12
• PGSA absolute scores over Baseline, Week 6 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pankovich, Study Director — BioWest Therapeutics Inc